CLINICAL TRIAL: NCT02555501
Title: Laser Therapy Associated With Photodynamic Therapy in the Treatment of Oral Mucositis Induced by Chemotherapy in Young Patients: Randomized Blind Clinical Trial
Brief Title: Oral Mucositis and Laser Therapy Associated With Photodynamic Therapy
Acronym: OMLTPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade Ceuma (Other)
Collaborators: Fundação de Amparo à Pesquisa e Desenvolvimento Científico do Maranhão (Unknown)
Responsible Party: Principal Investigator, Meire Coelho Ferreira, Matheus Coelho Bandeca, Universidade Ceuma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCCF-060264-AM
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Oral Mucositis
Keywords: children; cancer; stomatitis; clinical trial; laser therapy, low-level; methylene blue; photochemotherapy
MeSH Terms: conditions — Stomatitis; Neoplasms | interventions — 1-phenyl-3,3-dimethyltriazene; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PDT + Low level laser (Experimental): PDT (photosensitizer and low level laser) and low level laser
  Photosensitizer: aqueous solution of 0.005% methylene blue; Low level laser: infrared emitter laser unit with active medium AsGaAl (Gallium Arsenide and Aluminium) and red emitter with active medium InGaAlP (phosphide and Indium, Gallium and Potassium)
  Interventions: Other: PDT + Low level laser
- Low level laser (Active Comparator): Low level laser: infrared emitter laser unit with active medium AsGaAl (Gallium Arsenide and Aluminium) and red emitter with active medium InGaAlP (phosphide and Indium, Gallium and Potassium)
  Interventions: Radiation: Low level laser

INTERVENTIONS:
Other: PDT + Low level laser — Two days before the laser treatment, the side of the oral cavity chosen for the experimental treatment was pigmented with aqueous solution of 0.005% methylene blue. A ball of sterile cotton was soaked in the dye solution and placed in the center of the lesion. Photosensitizer remained in the place for 5 minutes (pre-irradiation period). Then, to activate the dye, the lesion was irradiated with red light (InGaAlP / phosphide and Indium, Gallium and potassium).
  From the 3rd to the 10th day was carried out only laser therapy. For laser therapy was first used infrared emitter laser unit with active medium AsGaAl (Gallium Arsenide and Aluminium). Then, we used the red emitter, whose active medium was the InGaAlP (phosphide and Indium, Gallium and Potassium).
  Arms: PDT + Low level laser
Radiation: Low level laser — Two days before the laser treatment, the lesion of the side of the oral cavity chosen for the control treatment was treated with ball of sterile cotton soaked in distilled water and the laser unit placed on the lesion without activation of the light. From the 3rd to the 10th day was carried out laser therapy. For laser therapy was first used infrared emitter laser unit with active medium AsGaAl (Gallium Arsenide and Aluminium). Then, we used the red emitter, whose active medium was the InGaAlP (phosphide and Indium, Gallium and Potassium).
  Arms: Low level laser

SUMMARY:
The aim of the study was to evaluate the therapeutic action through the diameter of the lesion, of low level laser (LLL) associated to photodynamic therapy (PDT) in oral mucositis (OM) lesions, in young patients. A randomized clinical trial blinded, split-mouth was performed. The study sample consisted of 15 cancer patients (3-16 years old) of Aldenora Bello Hospital (São Luís, Maranhão, Brazil). Random allocation by lot of treatments (PDT + LLL and LLL) to quadrants of the oral cavity was performed, and the patient was his own control. Patients were masked about therapy performed on each side of the arch. The evaluation period of both therapeutic regimens was 8 days, and the outcome assessed was the lesion size (measured in cm²). Friedman and Wilcoxon tests were applied and the effect magnitude calculated. The significance level was 5%. Statistically significant difference was observed between the groups for the lesion diameter of the 6th to the 8th day (greater regression of lesion size for the PDT + LLL group), which was confirmed by a difference magnitude moderated. Based on the findings, it is concluded that PDT + LLL showed greater therapeutic effect when compared to LLL in reducing the severity of OM lesions.

DETAILED DESCRIPTION:
The blind randomized clinical trial included 18 young patients, between 3 and 16 years old, undergoing chemotherapy or chemo/radiological the pediatric ward of Aldenora Bello Hospital in São Luís (Maranhão, Brazil). The study was conducted from October/2014 to January/2015. It was adopted as inclusion criteria patients between 3 and 18 years old, in the inductive phase of chemotherapy, with oral mucositis (OM) and bilateral lesions.

A mouth split model was conducted, and the patients were their own controls. The entry of the patients in the study occurred consecutively. To each patient, the operator/examiner drafted an envelope containing treatments to either side, being masked patient about the treatment of each side: PDT (photosensitized and low level laser) + low level laser; Low level laser].

The following parameters were used for the calculation of sample size: 95% confidence level, 80% statistical power and minimal difference of 0.82 point in the lesions diameter detected between paired samples. A "n" sample minimum of 14 was determined for each treatment. In order to compensate for possible losses, 18 patients were treated.

The treatments (PDT and low level laser; Low level laser) were performed in a hospital bed. Prior to treatment, the OM lesions were evaluated and a lesion on each side was chosen. Lesions should be located at the same site on both sides. The chosen site was the lip mucosa. Before the procedure, the patient was instructed as to brushing and not using mouthwashes, followed by cleaning of the oral cavity with gauze and distilled water. Two days before the laser treatment, the side of the oral cavity chosen for the experimental treatment (PDT and low level laser) was pigmented with the photosensitizer (aqueous solution of 0.005% methylene blue). A ball of sterile cotton was soaked in the dye solution and placed in the center of the lesion. Photosensitizer remained in the place for 5 minutes (pre-irradiation period). Then, to activate the dye, the lesion was irradiated with red light (InGaAlP / phosphide and Indium, Gallium and potassium) (Flash Laser III, DMC, São Carlos, São Paulo, Brazil), with a wavelength of 660 nm, for a period 90 seconds, with a power of 100mW, to 1cm away, according to the manufacturer's specifications. The lesion on the opposite side was treated with ball of sterile cotton soaked in distilled water and the laser unit placed on the lesion without activation of the light. This procedure aimed to mask the patient about the side that received the experimental therapy (PDT and low level laser). This masking was possible because the experimental solution is insipid, very soluble and thus leaves no residue.

From the 3rd to the 10th day (total of 8 days) was carried out only laser therapy on both sides. Lesions were evaluated until the 8th day. After the 8th day of assessment, the lesions were only treated to a complete remission as well as other lesions present in the oral cavity. For laser therapy was first used infrared emitter laser unit with active medium AsGaAl (Gallium Arsenide and Aluminium), with wavelength of 808nm, for analgesia. Then, the investigators used the red emitter, whose active medium was the InGaAlP (phosphide and Indium, Gallium and Potassium), with wavelength of 660nm to photobiomodulation. For both units emitting laser, the tip of the device was closed against the edges of the lesion, perpendicular to the tissue. A irradiation was continuous and the application punctual (10 seconds). The distance between the points of irradiation was about 1cm. The energy delivered was 4J per point of application. The interval between sessions was 24 hours.

The tip of the laser was disinfected with 70% alcohol solution and wrapped with a plastic film. Patients and operators wore glasses for eye protection.

A questionnaire containing demographic, socioeconomic and type of treatment for cancer was applied to parents and children. White blood cell count and platelets (beginning and end of the inductive phase of QT) were extracted from medical records.

The assessed outcome measure was the diameter of the lesion (in cm2). The areas of the lesions were measured with a flexible ruler (record made in cm2) by the operator/examiner from the start of treatment with exclusive laser therapy (3rd day). This procedure was repeated on subsequent days until the 8th day of laser treatment. The measurement of the lesions occurred prior to laser therapy applications.

The Friedman test was used for multiple comparisons within groups (different times of treatment). Paired evaluation between each two moments was evaluated using the Wilcoxon test, with significance corrected by Bonferroni test (p = 0.0071). The Wilcoxon test was used to compare the diameter of the lesion, every day, between the PDT + Low level laser and Low level laser groups (dependent samples/split-mouth). It calculated the effect magnitude (d) of standardized differences between averages of two groups. The level of significance for analysis was 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 3 and 18 years old
* Patients on chemotherapy inductive phase
* Patients with oral mucositis and bilateral lesions

Exclusion Criteria:

* Patients outside the established age
* Patients who are in other phases of chemotherapy
* Patients who did not have bilateral lesions

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Lesion size | 8 days
  Lesion size measured in cm²

CONTACTS AND LOCATIONS:
Overall Officials: Meire C. Ferreira, PhD, Study Director — Programa de Mestrado em Odontologia
Locations (1):
- Hospital Aldenora Bello, São Luís, Maranhão, Brazil

REFERENCES:
- [Background] Braga PE, Latorre Md Mdo R, Curado MP. [Childhood cancer: a comparative analysis of incidence, mortality, and survival in Goiania (Brazil) and other countries]. Cad Saude Publica. 2002 Jan-Feb;18(1):33-44. doi: 10.1590/s0102-311x2002000100004. Portuguese. PMID 11910422
- [Background] Instituto Nacional do Câncer (Brasil). Incidência de Câncer no Brasil: Estimativa 2014/2015. Rio de Janeiro: INCA, 2014.
- [Background] Bonan PRF, Lopes MA, Alves FA, Almeida OP. Clinical, biological, histopathological and proposed treatments for oral mucositis induced by radiation therapy: Literature Review. J Oncol 2005; 51:235-42.
- [Background] Sonis ST. Pathobiology of mucositis. Semin Oncol Nurs. 2004 Feb;20(1):11-5. doi: 10.1053/j.soncn.2003.10.003. PMID 15038512
- [Background] Chan KK, Oza AM, Siu LL. The statins as anticancer agents. Clin Cancer Res. 2003 Jan;9(1):10-9. PMID 12538446
- [Background] Reichart PA, Philipsen HP. Oral Pathology; Trad. John Peter Stein and Maximiano Ferreira Tovo. Porto Alegre: Medical Arts South; 2000.
- [Background] Andrade MC, Ribeiro AP, Dovigo LN, Brunetti IL, Giampaolo ET, Bagnato VS, Pavarina AC. Effect of different pre-irradiation times on curcumin-mediated photodynamic therapy against planktonic cultures and biofilms of Candida spp. Arch Oral Biol. 2013 Feb;58(2):200-10. doi: 10.1016/j.archoralbio.2012.10.011. Epub 2012 Nov 13. PMID 23153629
- [Background] Lee YH, Park HW, Lee JH, Seo HW, Lee SY. The photodynamic therapy on Streptococcus mutans biofilms using erythrosine and dental halogen curing unit. Int J Oral Sci. 2012 Dec;4(4):196-201. doi: 10.1038/ijos.2012.63. Epub 2012 Dec 7. PMID 23222991
- [Background] Mattiello FD, Coelho AA, Martins OP, Mattiello RD, Ferrao Junior JP. In vitro effect of photodynamic therapy on aggregatibacter actinomycetemcomitans and Streptococcus sanguinis. Braz Dent J. 2011;22(5):398-403. doi: 10.1590/s0103-64402011000500009. PMID 22011896
- [Background] Miyabe M, Junqueira JC, Costa AC, Jorge AO, Ribeiro MS, Feist IS. Effect of photodynamic therapy on clinical isolates of Staphylococcus spp. Braz Oral Res. 2011 May-Jun;25(3):230-4. doi: 10.1590/s1806-83242011005000006. Epub 2011 Feb 25. PMID 21359491
- [Background] Ishiyama K, Nakamura K, Ikai H, Kanno T, Kohno M, Sasaki K, Niwano Y. Bactericidal action of photogenerated singlet oxygen from photosensitizers used in plaque disclosing agents. PLoS One. 2012;7(5):e37871. doi: 10.1371/journal.pone.0037871. Epub 2012 May 22. PMID 22629466
- [Background] Corti L, Chiarion-Sileni V, Aversa S, Ponzoni A, D'Arcais R, Pagnutti S, Fiore D, Sotti G. Treatment of chemotherapy-induced oral mucositis with light-emitting diode. Photomed Laser Surg. 2006 Apr;24(2):207-13. doi: 10.1089/pho.2006.24.207. PMID 16706701
- [Background] Sonis ST. Mucosite oral em câncer de cabeça e pescoço: risco, biologia e gestão. Am Soc Clin Oncol Educ Book 2013; 33: 236.
- [Background] Sonis ST, Fazio RC, Fang L. Principles and Practice of Oral Medicine. 2 ed. Rio de Janeiro: Guanabara Koogan; 1996.
- [Background] Brown CG, Wingard J. Clinical consequences of oral mucositis. Semin Oncol Nurs. 2004 Feb;20(1):16-21. doi: 10.1053/j.soncn.2003.10.004. PMID 15038513
- [Background] Sonis ST. Mucositis as a biological process: a new hypothesis for the development of chemotherapy-induced stomatotoxicity. Oral Oncol. 1998 Jan;34(1):39-43. doi: 10.1016/s1368-8375(97)00053-5. PMID 9659518
- [Background] Cheng KK, Chang AM, Yuen MP. Prevention of oral mucositis in paediatric patients treated with chemotherapy; a randomised crossover trial comparing two protocols of oral care. Eur J Cancer. 2004 May;40(8):1208-16. doi: 10.1016/j.ejca.2003.10.023. PMID 15110885
- [Background] Hejna M, Kostler WJ, Raderer M, Steger GG, Brodowicz T, Scheithauer W, Wiltschke C, Zielinski CC. Decrease of duration and symptoms in chemotherapy-induced oral mucositis by topical GM-CSF: results of a prospective randomised trial. Eur J Cancer. 2001 Nov;37(16):1994-2002. doi: 10.1016/s0959-8049(01)00132-0. PMID 11597376
- [Background] Kostler WJ, Hejna M, Wenzel C, Zielinski CC. Oral mucositis complicating chemotherapy and/or radiotherapy: options for prevention and treatment. CA Cancer J Clin. 2001 Sep-Oct;51(5):290-315. doi: 10.3322/canjclin.51.5.290. PMID 11577493
- [Background] Martens LC. Laser physics and a review of laser applications in dentistry for children. Eur Arch Paediatr Dent. 2011 Apr;12(2):61-7. doi: 10.1007/BF03262781. PMID 21473835
- [Background] Costa AC, de Campos Rasteiro VM, Pereira CA, da Silva Hashimoto ES, Beltrame M Jr, Junqueira JC, Jorge AO. Susceptibility of Candida albicans and Candida dubliniensis to erythrosine- and LED-mediated photodynamic therapy. Arch Oral Biol. 2011 Nov;56(11):1299-305. doi: 10.1016/j.archoralbio.2011.05.013. Epub 2011 Jun 24. PMID 21704304
- [Background] Costa AC, Campos Rasteiro VM, da Silva Hashimoto ES, Araujo CF, Pereira CA, Junqueira JC, Jorge AO. Effect of erythrosine- and LED-mediated photodynamic therapy on buccal candidiasis infection of immunosuppressed mice and Candida albicans adherence to buccal epithelial cells. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Jul;114(1):67-74. doi: 10.1016/j.oooo.2012.02.002. Epub 2012 May 22. PMID 22727094
- [Result] Albuquerque ILS, Camargo TC. Prevention and Treatment of oral mucositis induced by radiation therapy: Literature Review. J Oncol 2007; 53:195-209.
- [Result] Lino MD, Carvalho FB, Oliveira LR, Magalhaes EB, Pinheiro AL, Ramalho LM. Laser phototherapy as a treatment for radiotherapy-induced oral mucositis. Braz Dent J. 2011;22(2):162-5. doi: 10.1590/s0103-64402011000200013. PMID 21537592
- [Result] Oberoi S, Zamperlini-Netto G, Beyene J, Treister NS, Sung L. Effect of prophylactic low level laser therapy on oral mucositis: a systematic review and meta-analysis. PLoS One. 2014 Sep 8;9(9):e107418. doi: 10.1371/journal.pone.0107418. eCollection 2014. PMID 25198431
- [Result] Carvalho PA, Jaguar GC, Pellizzon AC, Prado JD, Lopes RN, Alves FA. Evaluation of low-level laser therapy in the prevention and treatment of radiation-induced mucositis: a double-blind randomized study in head and neck cancer patients. Oral Oncol. 2011 Dec;47(12):1176-81. doi: 10.1016/j.oraloncology.2011.08.021. Epub 2011 Sep 10. PMID 21911312
- [Result] Figueiredo AL, Lins L, Cattony AC, Falcao AF. Laser therapy in the control of oral mucositis: a meta-analysis. Rev Assoc Med Bras (1992). 2013 Sep-Oct;59(5):467-74. doi: 10.1016/j.ramb.2013.08.003. Epub 2013 Oct 10. English, Portuguese. PMID 24119379
- [Result] Kharkwal GB, Sharma SK, Huang YY, Dai T, Hamblin MR. Photodynamic therapy for infections: clinical applications. Lasers Surg Med. 2011 Sep;43(7):755-67. doi: 10.1002/lsm.21080. PMID 22057503
- [Result] Cieplik F, Tabenski L, Buchalla W, Maisch T. Antimicrobial photodynamic therapy for inactivation of biofilms formed by oral key pathogens. Front Microbiol. 2014 Aug 12;5:405. doi: 10.3389/fmicb.2014.00405. eCollection 2014. PMID 25161649
- [Result] Abramoff MM, Lopes NN, Lopes LA, Dib LL, Guilherme A, Caran EM, Barreto AD, Lee ML, Petrilli AS. Low-level laser therapy in the prevention and treatment of chemotherapy-induced oral mucositis in young patients. Photomed Laser Surg. 2008 Aug;26(4):393-400. doi: 10.1089/pho.2007.2144. PMID 18754720
- [Result] Kuhn A, Porto FA, Miraglia P, Brunetto AL. Low-level infrared laser therapy in chemotherapy-induced oral mucositis: a randomized placebo-controlled trial in children. J Pediatr Hematol Oncol. 2009 Jan;31(1):33-7. doi: 10.1097/MPH.0b013e318192cb8e. PMID 19125084
- [Result] Bensadoun RJ, Franquin JC, Ciais G, Darcourt V, Schubert MM, Viot M, Dejou J, Tardieu C, Benezery K, Nguyen TD, Laudoyer Y, Dassonville O, Poissonnet G, Vallicioni J, Thyss A, Hamdi M, Chauvel P, Demard F. Low-energy He/Ne laser in the prevention of radiation-induced mucositis. A multicenter phase III randomized study in patients with head and neck cancer. Support Care Cancer. 1999 Jul;7(4):244-52. doi: 10.1007/s005200050256. PMID 10423050
- [Result] Sandoval RL, Koga DH, Buloto LS, Suzuki R, Dib LL. Management of chemo- and radiotherapy induced oral mucositis with low-energy laser: initial results of A.C. Camargo Hospital. J Appl Oral Sci. 2003 Dec;11(4):337-41. doi: 10.1590/s1678-77572003000400012. PMID 21394411
- [Result] Ferreira MVL, Sousa GR, Silveira LB, Amorim JCF. Aplicações da PDT - Terapia Fotodinâmica - na Clínica Odontológica. DMC Journal 2010; 6: 40-4.
- [Result] Cauwels RG, Martens LC. Low level laser therapy in oral mucositis: a pilot study. Eur Arch Paediatr Dent. 2011 Apr;12(2):118-23. doi: 10.1007/BF03262791. PMID 21473845
- [Result] Cruz LB, Ribeiro AS, Rech A, Rosa LG, Castro CG Jr, Brunetto AL. Influence of low-energy laser in the prevention of oral mucositis in children with cancer receiving chemotherapy. Pediatr Blood Cancer. 2007 Apr;48(4):435-40. doi: 10.1002/pbc.20943. PMID 16862549